CLINICAL TRIAL: NCT00082173
Title: Phase 2 Randomized Trial of a Moxifloxacin-Containing Regimen For Treatment of Smear-Positive Pulmonary Tuberculosis in Adults With and Without HIV Infection
Brief Title: Moxifloxacin As Part of a Multi-Drug Regimen For Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Dr. Richard E. Chaisson, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FD-R-002135-01
Record Dates: First submitted 2004-04-30; First posted 2004-05-04 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): INH 300mg/RIF 600mg/PZA 20mg/kg/MOX 400mg/EMB placebo once daily for 8 weeks
  Interventions: Drug: Moxifloxacin
- 2 (Placebo Comparator): INH 300mg/RIF 600mg/PZA 20mg/kg/MOX placebo/EMB 15-20mg/kg once daily for 8 weeks
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — 400mg daily for 8 weeks
  Other Names: Avelox

SUMMARY:
Current treatment of tuberculosis (TB) requires patients to take four drugs for 8 weeks and then two drugs for 4 months. New drug regimens that are shorter and effective against drug-resistant TB are needed. This study will evaluate whether using the drug moxifloxacin (MOX) in place of ethambutol (EMB) during the first 8 weeks of treatment will effectively treat TB.

DETAILED DESCRIPTION:
Approximately one-third of the world's population is infected with Mycoplasma tuberculosis; 7 to 8 million new cases of active TB occur each year. TB is the second most common infectious cause of death worldwide. Appropriate treatment of persons with active TB is very important in limiting the transmission of M. tuberculosis and preventing TB-related mortality. Current therapy requires 6 months of a four-drug regimen of isoniazid (INH), rifampin (RIF), pyrazinamide (PZA), and EMB.

The development of alternative regimens is a priority, and new classes of antituberculosis agents are needed to provide treatment options for patients with drug-resistant disease. This study will evaluate the effectiveness of replacing EMB with MOX in a multi-drug regimen in the initial phase of treatment of smear-positive pulmonary TB in patients with and without HIV infection.

Participants in this study will be randomly assigned to receive either a MOX-containing drug regimen or the standard EMB-containing drug regimen for 8 weeks. Participants will have study visits weekly during these 8 weeks. After 8 weeks, participants will discontinue MOX, EMB, and PZA and will continue taking INH and RFP for 4 months. Participants will have study visits at Months 4, 6, 12, and 18. Study visits will include a medical interview, physical exam, blood and urine tests, and sputum tests for TB.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive diagnosis of smear-positive pulmonary TB within 2 weeks of study entry. Patients with both pulmonary and extrapulmonary disease are eligible.
* Documentation of HIV infection status. If HIV status is unknown at study entry, the participant must consent to testing and results must be available prior to study participation.
* Agree to use acceptable methods of contraception

Exclusion Criteria:

* History of adverse drug reaction to MOX, INH, RIF, PZA, or EMB
* Disease or condition for which MOX, INH, RIF, PZA, or EMB is contraindicated
* History of more than 14 days of continuous antituberculosis therapy during the previous 2 years or more than 2 months of antituberculosis therapy ever
* Active AIDS-related opportunistic infection or malignancy
* Currently receiving or planning to receive HIV protease inhibitors or nonnucleoside reverse transcriptase inhibitors in the first 2 months after study entry
* Silicotuberculosis
* Central nervous system TB
* Pregnant or breastfeeding
* Unable to take oral medication
* Electrocardiogram (EKG) QTc interval greater than 450 msec
* Taking classes IA or III antiarrhythmic agents (quinidine, procainamide, amiodarone, sotalol), cisapride, erythromycin, perphenazine/amitriptyline, phenothiazines, or tricyclic antidepressant
* Diseases or conditions for which treatment with other drugs with antituberculosis activity (e.g., rifabutin for MAC prophylaxis) is anticipated during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Chaisson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Clementino Fraga Filho Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Conde MB, Efron A, Loredo C, De Souza GR, Graca NP, Cezar MC, Ram M, Chaudhary MA, Bishai WR, Kritski AL, Chaisson RE. Moxifloxacin versus ethambutol in the initial treatment of tuberculosis: a double-blind, randomised, controlled phase II trial. Lancet. 2009 Apr 4;373(9670):1183-9. doi: 10.1016/S0140-6736(09)60333-0. PMID 19345831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with respiratory symptoms suggestive of TB were recruited from the HUCFF outpatient TB clinic as well as other local TB clinics.
Pre-assignment Details: Patients who did not meet enrollment criteria or who did not want to participate in the study were excluded.
Groups:
- Experimental Arm: INH 300mg/RIF 600mg/PZA 20mg/kg/MOX 400mg/EMB placebo once daily for 8 weeks
- Control Arm: INH 300mg/RIF 600mg/PZA 20mg/kg/MOX placebo/EMB 15-20mg/kg once daily for 8 weeks
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started | 74 | 72
Completed | 64 | 61
Not Completed | 10 | 11
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Culture negative or resistant at baselin | 5 | 6

BASELINE CHARACTERISTICS:
Population: 125 had 8-week data (moxifloxacin n=64, ethambutol n=61)
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm (Moxi) | Control Arm (EMB) | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 71 | 143
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 32.5 (11.7) | 35.7 (12.0) | 34.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 22 | 56
  Male | 40 | 50 | 90
Region of Enrollment [Number; unit: participants]
  Brazil | 74 | 72 | 146

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Sterile Sputum Cultures
Description: Proportion of patients with sterile sputum cultures
Time Frame: 8 weeks
Population: Proportion of patients with sterile sputum cultures at week 8
Measure: Number; unit: Participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 64 | 61
Participants | 59 | 45

2. Secondary Outcome: Proportion of Patients With Grade 3 or 4 Adverse Reactions Attributable to Study Medications
Description: Proportion of patients with Grade 3 or 4 adverse reactions attributable to study medications
Time Frame: 8 weeks
Population: DAIDS Table of Adverse Events
Measure: Number; unit: Participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 74 | 72
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Experimental Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 6/74 | 6/72
Other Adverse Events (participants affected / at risk) | 0/74 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=74) | Control Arm (N=72)
Hospitalization (General disorders) | 3 (4) | 3 (3) — Hospitalization AEs for this study included:Community acquired pneumonia, abscess, D&C, edema and polyneuropathy, none related to study drugs
Death (Cardiac disorders) | 3 (3) | 5 (5) — Causes of deaths in the study included: sepsis, gunshots, neoplasm, intracranial hemorrhage, PTB and unknown, none related to study medications
Grade 4 event (Renal and urinary disorders) | 1 (1) | 0 (0) — Proteinuria, judged to be not related to study drugs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No